CLINICAL TRIAL: NCT05360290
Title: The Value of Circulating Tumor Cells in Patients With Breast Cancer Who Completed Surgery After Neoadjuvant Treatment: a Multicenter, Prospective Clinical Trial
Brief Title: CTCs in Breast Cancer After Neoadjuvant Treatment and Surgery: a Multicenter, Prospective Clinical Trial
Acronym: CTCNeoBC-E
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Wenjin Yin, Deputy Chief of Breast Surgery Department, RenJi Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: KY2022-044-B
Record Dates: First submitted 2022-04-23; First posted 2022-05-04 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Circulating Tumor Cell
MeSH Terms: conditions — Breast Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTC positive (Active Comparator)
  Interventions: Device: GILUPI CellCollector®
- CTC negative (Other)
  Interventions: Device: GILUPI CellCollector®

INTERVENTIONS:
Device: GILUPI CellCollector® — Use of GILUPI CellCollector® to detect CTC

SUMMARY:
The GILUPI CellCollector® is the first in vivo CTC isolation product worldwide, which is CE approved. This is a prospective, multicenter study to evaluate the prognostic value of circulating tumor cells in breast cancer patients who completed surgery after neoadjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged ≥18 and ≤70 years;
* Histologically confirmed invasive breast cancer (cT2-4N0-2M0 or cT1N1-3M0 before neoadjuvant treatment);
* Completed neoadjuvant treamtment and surgery (within 4 years after surgery);
* Administered neoadjuvant chemotherapy (regardless of chemotherapy regimen);
* ECOG 0-1

Exclusion Criteria:

* Metastatic disease (Stage IV);
* Female patients who are pregnancy or lactation;
* Uncontrollable puncture site infection or systemic infection;

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Estimated)
Dates: Start 2022-09-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
invasive disease-free survival (iDFS) | From surgery until time of event up to 3 years
  Invasive disease-free survival time is defined as the time from date of randomization until the first occurrence of invasive disease recurrence, distant metastasis and death from any cause.

SECONDARY OUTCOMES:
pathological complete response (pCR) | at surgery
  ypT0 ypN0, ypT0/is ypN0, ypT0 or ypT0/is
overall Survival (OS) | From surgery until time of event up to 3 years
  Overall survival is defined as the time from randomization to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided